CLINICAL TRIAL: NCT02178397
Title: A Multicenter Randomized Phase III Study Comparing Second-line Treatment With Chemotherapy Associated or Not to Erlotinib in NSCLC Patients With Secondary Resistance to TKI-EGFR
Acronym: FLARE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: Centre Francois Baclesse (Other)
Collaborators: Groupe Francais De Pneumo-Cancerologie (Other); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FLARE /GFPC 03-2013
Record Dates: First submitted 2014-06-25; First posted 2014-06-30 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2016-07

CONDITIONS: NSCLC Patients With EGFR Activating Mutation
Keywords: erlotinib; lung cancer; EGFR mutation
MeSH Terms: conditions — Lung Neoplasms | interventions — Erlotinib Hydrochloride; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EXPERIMENTAL ARM B (Experimental): INDUCTION chemotherapy: 4 cycles of
  * pemetrexed with cisplatin or carboplatin
  * or gemcitabine with cisplatin or carboplatin in combination with erlotinib
  THEN, for responders and for patients with stable disease :MAINTENANCE chemotherapy by Pemetrexed in combination with erlotinib
  Interventions: Drug: ERLOTINIB WITH CHEMOTHERAPY
- STANDARD ARM A (Active Comparator): INDUCTION chemotherapy: 4 cycles of
  * pemetrexed with cisplatin or carboplatin
  * or gemcitabine with cisplatin or carboplatin
  THEN, for responders and for patients with stable disease :MAINTENANCE chemotherapy by Pemetrexed
  Interventions: Drug: CHEMOTHERAPY ONLY

INTERVENTIONS:
Drug: ERLOTINIB WITH CHEMOTHERAPY
  Arms: EXPERIMENTAL ARM B
Drug: CHEMOTHERAPY ONLY
  Arms: STANDARD ARM A

SUMMARY:
The current first line treatment of patients with EGFR activating mutation lung cancer is EGFR TKI. Compared to platinum-based chemotherapy, EGFR-TKIs are superior in terms of response rate and progression-free survival. However, an acquired resistance occurs almost constantly. The second-line treatment includes platinum-based chemotherapy in the absence of contraindication. This chemotherapy is then administered after discontinuing EGFR TKIs.

However, a rebound phenomenon of the disease was described in patients who discontinued EGFR TKIs. Some clinical teams therefore recommend, as a precaution, in order to avoid any withdrawal phenomenon, to never discontinue EGFR TKIs in patients developing an EGFR TKI acquired resistance.

It seems therefore useful to conduct a study to better define the therapeutic strategy to adopt in patients developing an acquired resistance after having received EGFR TKIs as first line treatment.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged 18 years or more
* Non-small cell lung cancer carcinoma (NSCLC) cytologically or histologically confirmed
* Measurable disease according to RECIST 1.1 criteria
* Life expectancy greater than 12 weeks
* Performance Status (ECOG) ≤ 2
* Stage IIIB considered ineligible for thoracic radiotherapy at "curative" doses or stage IV
* Presence of at least one measurable target lesion
* Documented disease progression (RECIST 1.1) after first line treatment with erlotinib, during at least 4 months in case of partial or complete response according to RECIST criteria, or 6 months in case of stable disease. The treatment with Erlotinib should not be discontinued for more than 8 days between the progression and the inclusion in the study. The daily dose of Erlotinib should be at least 50 mg.
* Presence of one of the EGFR activating mutations in the tumor (exon 19 deletion or L858R, G719X or L861Q)
* One additional line of previous chemotherapy is allowed if administered in adjuvant or neoadjuvant setting and received more than six months before.
* Prior radiotherapy is allowed if the volume of irradiated marrow is <25% of the total bone marrow. The prior radiotherapy must be completed at least two weeks before study entry
* Brain metastases are allowed if they are controlled without steroids and if their treatment is completed (radiotherapy and/or surgery). Patients with no symptomatic brain metastases may be included; even if brain metastases are progressive and even if they are the only site of progression (since the investigator considers that irradiation is not required). These metastases have not to be life-threatening (are excluded: cerebellar metastasis ≥ 2 cm, brainstem metastasis, brain metastasis > 3 cm and/or near important functional structure).
* Normal Liver function (bilirubin ≤ULN, AST - ALT ≤2.5 x ULN, alkaline phosphatase ≤3 x ULN), or in case of liver metastases: alkaline phosphatase, AST-ALT ≤ 5 x ULN
* Normal renal function: blood creatinine ≤ULN and / or creatinine clearance> 60 ml/min calculated with the MDRD formula
* Normal blood function: absolute neutrophil count ≥ 1.5 x 109/l and / or platelets ≥ 100 x 109 / l, hemoglobin> 9 g/dl
* Woman and man under efficient contraception during treatment and at least 6 months after the end of treatment by pemetrexed or platinum or gemcitabine
* Signed written Informed consent

Exclusion Criteria:

* Bronchoalveolar, mixed, neuroendocrine and small cell lung cancers
* Patient with only bone metastases are not eligible
* All progressive metastatic sites treated locally (surgery, radiotherapy)
* Superior vena cava syndrome
* Uncontrolled cardiac disease requiring treatment
* Congestive heart failure, angina pectoris, significant arrhythmias or history of myocardial infarction within the previous 12 months
* Neurological or psychiatric disorders
* Uncontrolled infectious disease
* Peripheral neuropathy grade≥ 2
* Definitive contraindication for the use of steroids
* Inductive anti-epileptic treatments (phenobarbital, phenytoïne)• Previous or concomitant other cancer, including skin cancer (except basal cell cancer of the skin), except in situ treated carcinoma of the cervix , except cancer treated with surgery alone without recurrence for 5 years
* Pregnant or breastfeeding woman
* Patient follow-up not achievable
* Participation in a trial within the last 30 days
* Patient deprived of liberty as a result of a justice or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Efficacy by PFS | From date of randomization until the date of first documented progression evaluated every 6-9 weeks
  Efficacy will be assessed by the PFS, define as time between randomization of the patient in the study and disease progression (local, regional, distant and second cancer) or death (all causes). Alive patients free of progression will be censored at the last follow-up.

SECONDARY OUTCOMES:
scores of QoL | at 4 months after inclusion
  difference between the scores of QoL at baseline and at 4 months after inclusion for the three targeted dimensions of EORTC QLQ-C30 (global quality of life, fatigue and physical functioning). A difference or 10 points or more at 4 months after inclusion for one score between the 2 arms will be considered as clinically relevant.
Overall survival | From date of randomization until the date of death from any cause, whichever came first, assessed up to 100 months
  Overall survival defined as time interval between randomization and death (all causes). Alive patients will be censored at the last date of news or data cut off
Tumoral response | every 6-9 weeks
  Tumoral response (complete response, partial response, stable disease, progression) according to RECIST 1.1
Toxicities | From date of randomization until study participation, assessed up to 100 months
  Toxicities according to NCI-CTC-AE v.4
Rebound phenomenon (flare) | within 3 weeks after disease progression before inclusion
  Rebound phenomenon (flare) defined by a hospitalization or a death within 3 weeks for disease progression after the end of TKI EGFR treatment (in the arm without EGFR TKI) and date of onset

CONTACTS AND LOCATIONS:
Overall Officials: Radj GERVAIS, MD, Principal Investigator — Centre François Baclesse - CAEN- FRANCE
Locations (35):
- France (35):
  - CH, Aix-en-Provence
  - CH, Amiens
  - CHRU, Angers
  - CH, Annecy
  - CHU, Brest
  - Centre François BACLESSE, Caen
  - CHIC, Créteil
  - CH, Draguignan
  - CH, Elbeuf
  - CHIC, Gap
  - Ch La Roche/Yon, La Roche/yon
  - Centre Hospitalier, Le Mans
  - Centre Oscar Lambret, Lille
  - CHU, Limoges
  - CH, Longjumeau
  - CH, Lorient
  - CH, Mantes-la-Jolie
  - Institut Paoli Calmettes, Marseille
  - AP-HM - Hôpital Nord, Marseille
  - CH, Mâcon
  - CH, Meaux
  - Centre Hospitalier Intercommunal, Meulan-en-Yvelines
  - CH, Pau
  - Centre Catalan, Perpignan
  - CHU, Rennes
  - CH, Roanne
  - CHU, Rouen
  - CH, Saint-Brieuc
  - Institut de Cancérologie de la Loire, Saint-Etienne
  - CH, Salon-de-Provence
  - CH, Sens
  - Centre Paul Strauss, Strasbourg
  - CH, Tarbes
  - Hôpital d'instruction des Armées Sainte-Anne, Toulon
  - CH, Villefranche